CLINICAL TRIAL: NCT05725187
Title: Prospective Validation Study of Artificial Intelligence-based Prediction Algorithm for the Prediction of Paroxysmal Atrial Fibrillation
Brief Title: Prospective Validation Study of AI-based Prediction Algorithm for the Prediction of Paroxysmal Atrial Fibrillation
Acronym: PROVISION-AF
Status: Enrolling by invitation | Type: Observational
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Collaborators: Ewha Womans University Seoul Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROVISION-AF
Record Dates: First submitted 2023-01-20; First posted 2023-02-13 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: artificial intelligence; electrocardiogram
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Low risk group for paroxysmal atrial fibrillation: Subject patients are above 20 in age who are hospitalized in our hospital or outpatients with arrhythmia symptoms after the clinical research approval. The sinus rhythm electrocardiogram at the time of the patient's participation in the study is put into the artificial intelligence prediction algorithm, and the risk stratification results are blinded and are not informed to both the research director and the subjects. For the low-risk group, after attaching the wearable electrocardiogram to the subject, the electrocardiogram recorded a week later is analyzed to confirm the occurrence of atrial fibrillation.
  Interventions: Device: MobiCare
- High risk group for paroxysmal atrial fibrillation: Subject patients are above 20 in age who are hospitalized in our hospital or outpatients with arrhythmia symptoms after the clinical research approval. The sinus rhythm electrocardiogram at the time of the patient's participation in the study is put into the artificial intelligence prediction algorithm, and the risk stratification results are blinded and are not informed to both the research director and the subjects. For the highrisk group, after attaching the wearable electrocardiogram to the subject, the electrocardiogram recorded a week later is analyzed to confirm the occurrence of atrial fibrillation.
  Interventions: Device: MobiCare

INTERVENTIONS:
Device: MobiCare — It is a 9.2g wearable electrocardiogram device, mobiCARE, in the form of a patch, and the model name is MC200M.

SUMMARY:
The purpose of this study is to predict the occurrence of paroxysmal atrial fibrillation by finding high-risk group from normal sinus rhythm ECG through artificial intelligence-based prediction algorithm.

DETAILED DESCRIPTION:
This study is a multi-center, prospective observational validation study. Patients aged 18 or above who are hospitalized at our hospital or who visited the outpatient clinic with arrhythmia symptoms (such as palpitation) after the clinical research approval will be enrolled. The normal sinus rhythm electrocardiogram (ECG) at the time of participation in the study is recorded and put into the artificial intelligence prediction algorithm. The result of risk stratification is blinded and will not be informed to both the research director and subjects. After applying wearable devices to the subject, the ECG recorded for the first week is analyzed to confirm the occurrence of paroxysmal atrial fibrillation (the gold standard for diagnosis of atrial fibrillation). When the wearable devices are removed, the 12 lead electrocardiogram will be taken again, and if it shows normal sinus rhythm electrocardiogram, then it will be put into the artificial intelligence prediction algorithm to calculate the result as well.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be above 20 in age
* Participants are patients with symptom of arrhythmia who visited outpatient clinic or who have been hospitalized

Exclusion Criteria:

* Excluding patients with cardiac implantable electronic device such as pacemakers, implantable defibrillators (ICD), or cardiac resynchronization therapy (CRT).
* Excluding pregnant women and lactating women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are selected from adults above age of 20 with their consent with a target for patients who come to the hospital with arrhythmia symptoms from an outpatient clinic or who are admitted to a hospital.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of paroxysmal AF | 1 week
  The AI prediction algorithm classifies patients into high-risk and low-risk categories for predicting paroxysmal atrial fibrillation within a week, based on ECG recordings of those with normal sinus rhythm. The accuracy of the prediction will be assessed through the use of a wearable device that records occurrence of paroxysmal atrial fibrillation over the course of a week.

SECONDARY OUTCOMES:
Performance verification of AI prediction model | 1 week
  The artificial intelligence prediction algorithm categorizes patients into high-risk and low-risk groups when predicting paroxysmal atrial fibrillation within one week based on normal sinus rhythm ECG data. The AI prediction algorithm's performance is assessed based on the data obtained from the primary outcome, which involves confirming whether atrial fibrillation recorded through a week-long use of a wearable device. We will gauge the algorithm's effectiveness by evaluating its predictive abilities, encompassing sensitivity, specificity, positive predictive rate, negative predictive rate, and the F1 score.

OTHER OUTCOMES:
Predictive capabilities of AI prediction model compared to expert cardiologists | 10 minute
  The predictive capabilities of the artificial intelligence prediction algorithm in risk stratification will be compared to the risk stratification proficiency of the experts. Each expert will be required to answer a questionnaire consisting of 30 ECGs to classify them as high risk or low risk. The questionnaire is composed of three components:
  Q1. Atrial fibrillation/flutter risk prediction based on normal sinus rhythm 12-lead ECG and participant's clinical data (Age, gender, comorbidities, laboratory result, EHRA Symptom Score, etc.). The laboratory result could include BUN/Cr, eGFR, liver function test, lipid profile test.
  Q2. Further plan required for identification of atrial fibrillation/flutter. Q3. Decisive evidence of atrial fibrillation/flutter risk prediction. The evidence could include normal sinus rhythm 12-lead ECG or participant's clinical data.

CONTACTS AND LOCATIONS:
Overall Officials: Sumi Jung, Study Director — Ewha Womans University Mokdong Hospital
Locations (11):
- South Korea (11):
  - Chonnam National University Hospital, Gwangju
  - Yongin Severance Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Chungbuk National University Hospital, Jungbuk
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ribeiro AH, Ribeiro MH, Paixao GMM, Oliveira DM, Gomes PR, Canazart JA, Ferreira MPS, Andersson CR, Macfarlane PW, Meira W Jr, Schon TB, Ribeiro ALP. Automatic diagnosis of the 12-lead ECG using a deep neural network. Nat Commun. 2020 Apr 9;11(1):1760. doi: 10.1038/s41467-020-15432-4. PMID 32273514
- [Background] Willems S, Borof K, Brandes A, Breithardt G, Camm AJ, Crijns HJGM, Eckardt L, Gessler N, Goette A, Haegeli LM, Heidbuchel H, Kautzner J, Ng GA, Schnabel RB, Suling A, Szumowski L, Themistoclakis S, Vardas P, van Gelder IC, Wegscheider K, Kirchhof P. Systematic, early rhythm control strategy for atrial fibrillation in patients with or without symptoms: the EAST-AFNET 4 trial. Eur Heart J. 2022 Mar 21;43(12):1219-1230. doi: 10.1093/eurheartj/ehab593. PMID 34447995
- [Background] Park J, Shim J, Lee JM, Park JK, Heo J, Chang Y, Song TJ, Kim DH, Lee HA, Yu HT, Kim TH, Uhm JS, Kim YD, Nam HS, Joung B, Lee MH, Heo JH, Pak HN; RAFAS Investigators*. Risks and Benefits of Early Rhythm Control in Patients With Acute Strokes and Atrial Fibrillation: A Multicenter, Prospective, Randomized Study (the RAFAS Trial). J Am Heart Assoc. 2022 Feb;11(3):e023391. doi: 10.1161/JAHA.121.023391. Epub 2022 Jan 19. PMID 35043663
- [Background] Noseworthy PA, Attia ZI, Behnken EM, Giblon RE, Bews KA, Liu S, Gosse TA, Linn ZD, Deng Y, Yin J, Gersh BJ, Graff-Radford J, Rabinstein AA, Siontis KC, Friedman PA, Yao X. Artificial intelligence-guided screening for atrial fibrillation using electrocardiogram during sinus rhythm: a prospective non-randomised interventional trial. Lancet. 2022 Oct 8;400(10359):1206-1212. doi: 10.1016/S0140-6736(22)01637-3. Epub 2022 Sep 27. PMID 36179758
- [Background] Attia ZI, Noseworthy PA, Lopez-Jimenez F, Asirvatham SJ, Deshmukh AJ, Gersh BJ, Carter RE, Yao X, Rabinstein AA, Erickson BJ, Kapa S, Friedman PA. An artificial intelligence-enabled ECG algorithm for the identification of patients with atrial fibrillation during sinus rhythm: a retrospective analysis of outcome prediction. Lancet. 2019 Sep 7;394(10201):861-867. doi: 10.1016/S0140-6736(19)31721-0. Epub 2019 Aug 1. PMID 31378392